CLINICAL TRIAL: NCT02552706
Title: The Efficacy and Mechanisms of Oral Probiotics in Preventing Necrotizing Enterocolitis Among Very Low Birth Weight Infants With Formula-feeding
Brief Title: The Efficacy and Mechanisms of Oral Probiotics in Preventing Necrotizing Enterocolitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Bao'an Maternal and Child Health Hospital (Other)
Collaborators: China Medical University Hospital (Other); Shenzhen People's Hospital (Other); Shenzhen Sixth People's Hospital (Other); Longhua Hospital Of Baoan District, Shenzhen (Other)
Responsible Party: Principal Investigator, liyuefeng, Ward chief of department of neonatology, Shenzhen Bao'an Maternal and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LL2014006
Record Dates: First submitted 2015-09-12; First posted 2015-09-17 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2015-09

CONDITIONS: Necrotizing Enterocolitis; Death
Keywords: probiotics; preterm very low birth weight infants; necrotizing enterocolitis; gut microflora; TLR; NF-KB; inflammatory factors
MeSH Terms: conditions — Enterocolitis, Necrotizing; Death | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotics group (Experimental): Administration of probiotics 500mg begins by mouth within 4 hours of life with 1-3 consecutive doses; the frequency depends on the feeding times. Study is continuous until preterm infants grow up to 36 weeks post menstrual age.
  Interventions: Dietary Supplement: probiotics
- control group (Placebo Comparator): control group received 1 mL of a 5% glucose solution. Administration of control group begins by mouth within 4 hours of life with 1-3 consecutive doses; the frequency depends on the feeding times. Study is also continuous until preterm infants grow up to 36 weeks post menstrual age.
  Interventions: Dietary Supplement: glucose solution

INTERVENTIONS:
Dietary Supplement: probiotics — Administration of mixture probiotics 500mg by mouth, one time or divided into 2-4 times depends on the feeding volume until to 36 weeks post menstrual age.
  Arms: probiotics group
Dietary Supplement: glucose solution — Administration of 1 mL of a 5% glucose solution by mouth, one time or divided into 2-4 times depends on the feeding volume until to 36 weeks post menstrual age.
  Arms: control group

SUMMARY:
The purpose of this study is to investigate the efficacy and its mechanisms of oral mixture probiotics in preventing necrotizing enterocolitis among the preterm very low birth weight infants.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) remains the most catastrophic gastrointestinal emergencies in preterm very low birth weight (VLBW) infants.Although study showed it is a multifactorial disease, its pathogenesis is still not yet unclear currently. Prematurity and formula feeding is considered as the main risk factors.Gut microbiota disturbance and immature immune system is associated with NEC. A lot of studies had showed that oral probiotics can alter gut microbiota flora colonization and reduce the incidence of NEC,but the exact mechanism remains unclear.The aim of this study is to elucidate the clinical efficacy and possible molecular mechanism of oral mixture probiotics in preventing NEC among preterm VLBW infants.

Patient Registry procedures: First,randomized numbers was generated by the computer and sent to the principal investigator(PI) at each center when an infant was eligible for enrollment.Second, patient will be assigned randomly to experimental group or control group by PI.Finally,the PI at each center will be responsible for the accuracy,completeness or representativeness of medical records, registry forms,data collection.

Sample size determination: The incidence of death and NEC was around 20% recently.To reduce the incidence of NEC and death to 10% at discharge would require a 50% improvement.At 80% power at P = 0.05 (two-sided),the loss rate of 0.2, this would require 135 subjects per arm.

Statistical analysis:The two groups were compared by a Χ2-test for categorical variables,Mann-Whitney U Test were used when reporting medians.A P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ≦ 34 weeks gestational age and birth weight below 1500 gm and who survive to NICU are eligible for the trial.

Exclusion Criteria:

* severe asphyxia (stage III),
* fetal chromosomal anomalies,
* cyanotic congenital heart disease,
* congenital intestinal atresia, gastroschisis, omphalocele, active upper gastric intestinal bleeding,
* lacking/refused of parental consent,
* those who are fasted for >3 weeks during the study period.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
the incidence of combined death and necrotizing enterocolitis | at 36 weeks correct gestational age

SECONDARY OUTCOMES:
the incidence of sepsis,intraventricular hemorrhage(IVH)(grade 3-4),feeding intolerance(FI),bronchopulmonary dysplasia(BPD),parenteral nutrition associated liver disease(PNALD)and retinopathyof prematurity(ROP). | participants will be followed for the duration of hospital stay, an expected average of 8 weeks

OTHER OUTCOMES:
the influence of oral probiotics on gut microbiota and immunomodulatory | at birth, 2 and 4 weeks of life, 36 week correct gestational age.
  test fecal microbiota via high throughput sequencing and blood toll like receptor(TLR)2,TLR4,neclear factor kappa B(NF-KB)were detected using flow cytomtry.Inflammatory factors of blood were tested via Cytometric Bead Array(CBA).All above samples were obtained only from Shenzhen Bao'an Maternal and Child Health Hospital.The fecal DNA were first extracted at centre laboratory in aboved hospital and sent them to Beijing Genomics Institute(BGI) for further sequenceing ,if necessary, quantitative polymerase chain reaction(qPCR)of gut dominant bacterias related to late onset sepsis(LOS) will be tested for assessing the effect of oral probiotics on gut microbiota and underlying the mechanism. Flow cytometry analysis of TLR2,TLR4 and NF-KB were made by the senior laboratorian of our department and resposible for the accuracy of experimental result. CBA of inflammatory factors will be made by senting the blood samples to Beijing JIAMAY BIOLAB.

CONTACTS AND LOCATIONS:
Overall Officials: Yuefeng Li, M.D., Principal Investigator — Shenzhen Bao'an Maternal and Child Health Hospital; HungChih Lin, M.D., Study Director — China Medical University Hospital; Benqing Wu, M.D., Study Director — Shenzhen People's Hospital; Xiaodong Li, M.D., Study Director — Shenzhen Sixth People's Hospital; Zhangxin Wang, M.D., Study Director — Longhua Hospital Of Baoan District, Shenzhen
Locations (4):
- China (4):
  - Longhua People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Shenzhen Bao'an Maternal and Child Health Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Shenzhen Sixth People's Hospital, Shenzhen, Guangdong

REFERENCES:
- [Background] Lin HC, Hsu CH, Chen HL, Chung MY, Hsu JF, Lien RI, Tsao LY, Chen CH, Su BH. Oral probiotics prevent necrotizing enterocolitis in very low birth weight preterm infants: a multicenter, randomized, controlled trial. Pediatrics. 2008 Oct;122(4):693-700. doi: 10.1542/peds.2007-3007. PMID 18829790
- [Result] Genzel-Boroviczeny O, MacWilliams S, Von Poblotzki M, Zoppelli L. Mortality and major morbidity in premature infants less than 31 weeks gestational age in the decade after introduction of surfactant. Acta Obstet Gynecol Scand. 2006;85(1):68-73. doi: 10.1080/00016340500290947. PMID 16521683
- [Result] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Result] Rees CM, Pierro A, Eaton S. Neurodevelopmental outcomes of neonates with medically and surgically treated necrotizing enterocolitis. Arch Dis Child Fetal Neonatal Ed. 2007 May;92(3):F193-8. doi: 10.1136/adc.2006.099929. Epub 2006 Sep 19. PMID 16984980
- [Result] Huda S, Chaudhery S, Ibrahim H, Pramanik A. Neonatal necrotizing enterocolitis: Clinical challenges, pathophysiology and management. Pathophysiology. 2014 Feb;21(1):3-12. doi: 10.1016/j.pathophys.2013.11.009. Epub 2014 Feb 11. PMID 24525171
- [Result] Hall NJ, Eaton S, Pierro A. Royal Australasia of Surgeons Guest Lecture. Necrotizing enterocolitis: prevention, treatment, and outcome. J Pediatr Surg. 2013 Dec;48(12):2359-67. doi: 10.1016/j.jpedsurg.2013.08.006. PMID 24314171
- [Result] Quigley MA, Henderson G, Anthony MY, McGuire W. Formula milk versus donor breast milk for feeding preterm or low birth weight infants. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD002971. doi: 10.1002/14651858.CD002971.pub2. PMID 17943776
- [Result] Mshvildadze M, Neu J, Mai V. Intestinal microbiota development in the premature neonate: establishment of a lasting commensal relationship? Nutr Rev. 2008 Nov;66(11):658-63. doi: 10.1111/j.1753-4887.2008.00119.x. PMID 19019028
- [Result] Sharma R, Tepas JJ 3rd, Hudak ML, Mollitt DL, Wludyka PS, Teng RJ, Premachandra BR. Neonatal gut barrier and multiple organ failure: role of endotoxin and proinflammatory cytokines in sepsis and necrotizing enterocolitis. J Pediatr Surg. 2007 Mar;42(3):454-61. doi: 10.1016/j.jpedsurg.2006.10.038. PMID 17336180
- [Result] Nair V, Soraisham AS. Probiotics and prebiotics: role in prevention of nosocomial sepsis in preterm infants. Int J Pediatr. 2013;2013:874726. doi: 10.1155/2013/874726. Epub 2013 Jan 14. PMID 23401695
- [Result] Sarowska J, Choroszy-Krol I, Regulska-Ilow B, Frej-Madrzak M, Jama-Kmiecik A. The therapeutic effect of probiotic bacteria on gastrointestinal diseases. Adv Clin Exp Med. 2013 Sep-Oct;22(5):759-66. PMID 24285463
- [Result] Di Gioia D, Aloisio I, Mazzola G, Biavati B. Bifidobacteria: their impact on gut microbiota composition and their applications as probiotics in infants. Appl Microbiol Biotechnol. 2014 Jan;98(2):563-77. doi: 10.1007/s00253-013-5405-9. Epub 2013 Nov 28. PMID 24287935
- [Result] Liu Y, Fatheree NY, Mangalat N, Rhoads JM. Lactobacillus reuteri strains reduce incidence and severity of experimental necrotizing enterocolitis via modulation of TLR4 and NF-kappaB signaling in the intestine. Am J Physiol Gastrointest Liver Physiol. 2012 Mar 15;302(6):G608-17. doi: 10.1152/ajpgi.00266.2011. Epub 2011 Dec 29. PMID 22207578
- [Result] Deshpande G, Rao S, Patole S, Bulsara M. Updated meta-analysis of probiotics for preventing necrotizing enterocolitis in preterm neonates. Pediatrics. 2010 May;125(5):921-30. doi: 10.1542/peds.2009-1301. Epub 2010 Apr 19. PMID 20403939
- [Result] Lu P, Sodhi CP, Hackam DJ. Toll-like receptor regulation of intestinal development and inflammation in the pathogenesis of necrotizing enterocolitis. Pathophysiology. 2014 Feb;21(1):81-93. doi: 10.1016/j.pathophys.2013.11.007. Epub 2013 Dec 22. PMID 24365655
- [Result] Hackam DJ, Afrazi A, Good M, Sodhi CP. Innate immune signaling in the pathogenesis of necrotizing enterocolitis. Clin Dev Immunol. 2013;2013:475415. doi: 10.1155/2013/475415. Epub 2013 May 23. PMID 23762089
- [Result] Ganguli K, Meng D, Rautava S, Lu L, Walker WA, Nanthakumar N. Probiotics prevent necrotizing enterocolitis by modulating enterocyte genes that regulate innate immune-mediated inflammation. Am J Physiol Gastrointest Liver Physiol. 2013 Jan 15;304(2):G132-41. doi: 10.1152/ajpgi.00142.2012. Epub 2012 Nov 8. PMID 23139215
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2023 Jul 26;7(7):CD005496. doi: 10.1002/14651858.CD005496.pub6. PMID 37493095
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2020 Oct 15;10(10):CD005496. doi: 10.1002/14651858.CD005496.pub5. PMID 33058137